CLINICAL TRIAL: NCT02250547
Title: Optimization With SonR Method in the ClinicAl pRactice
Acronym: OSCAR
Status: Completed | Type: Observational
Sponsor: LivaNova (Industry)
Responsible Party: Sponsor
Other Study IDs: RCSY01 OSCAR
Record Dates: First submitted 2013-07-10; First posted 2014-09-26 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: CRT Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Evaluate the percentage of patients optimized at least once every month by the SonR automatic optimization method, until M6 follow-up, in Heart failure (HF) patients prevalently in sinus rhythm

DETAILED DESCRIPTION:
Thanks to the SonR technology it is possible to adjust the optimal VV and AV delays over time, in a fully automatic, time saving and operator independent way. It is possible to optimize the VV and AV delays in office, during follow-up visits, but also enable the automatic optimization that weekly optimize the AV and VV delays.

For the reasons mentioned above, the sponsor expects that the SonR optimization method increases the number of patients optimized systematically at each follow-up The purpose of this study is to evaluate the percentage of patients optimized at least once every month by the SonR automatic optimization method, until M6 follow-up, in HF patients prevalently in sinus rhythm.

The primary objective will be evaluated as the percentage of patients successfully optimized every month until M6.

A patient is considered successfully optimized by the SonR during one month if at least one Atri-Ventricular (AV) or Ventricular-Ventricular (VV) optimization is completed by the SonR automatic optimization method during the month.

Patients eligible for the analysis are those with SonR automatic optimization function enabled and at least 50% of the time in sinus rhythm

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible for implantation or implanted for less than 6 weeks (primo-implant, replacement, upgrade) with a a Paradym RF SonR CRT-D and SonRtip Atrial Lead, according to current available guidelines (RF=radio frequency)
* Patient has signed and dated informed consent (according to the laws and regulations of the country in which the observation is performed)

Exclusion Criteria:

* Persistent atrial arrhythmias
* Already included in another interventional clinical study
* Not available for routine follow-up visits
* Inability to understand the purpose of the study
* Under guardianship
* Under18 years old
* Drug addiction or abuse
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac resyncronisation therapy - defibrillator (CRT-D) patients
Sampling Method: Non-Probability Sample
Enrollment: 278 (Estimated)
Dates: Start 2012-07 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
evaluate the percentage of patients optimized at least once every month by the SonR automatic optimization method, until M6 follow-up, in HF patients prevalently in sinus rhythm | 6 months
  The primary objective will be evaluated as the percentage of patients successfully optimized every month until M6.
  A patient is considered successfully optimized by the SonR during one month if at least one AV or VV optimization is completed by the SonR automatic optimization method during the month.
  Patients eligible for the analysis are those with SonR automatic optimization function enabled and at least 50% of the time in sinus rhythm

SECONDARY OUTCOMES:
Percentage of patients with SonR automatic optimization function enabled at each follow-up | 6M
  The number of patients with automatic SonR optimization enabled over the total number of patients at: Implantation, Baseline, M6
Analyze the evolution of optimal AV and VV delays SonR optimized over time | 6M
  Compare the mean and the intra-patient AV and VV delays between consecutive follow-ups
Report system-related complications | 6M
  Report system-related complications

CONTACTS AND LOCATIONS:
Overall Officials: Carsten W Israel, Principal Investigator — Evangelischen Krankenhaus Bielefeld - Germany
Locations (21):
- Allgemeines Krankenhaus Linz (AKH LINZ), Linz, Austria
- France (12):
  - CH Sud Francilien, Corbeil Essonne
  - Centre Hospitalier de Haguenau, Haguenau
  - CH de Marne la Vallée, Jossigny
  - CMC du Mans - Pôle Santé Sud, Le Mans
  - Polyclinique du Bois, Lille
  - Chu Dupuytren, Limoges
  - CH St Philibert, Lomme
  - CH St Joseph et St Luc, Lyon
  - Polyclinique Beauregard, Marseille
  - Centre hospitalier Belford Montbéliard, Montbéliard
  - CH Poitiers, Poitiers
  - Hôpital Victor Provo, Roubaix
- Germany (2):
  - Evangelisches Krankenhaus, Bielefeld
  - PAP2 - Kardiologische Praxis Papenburg, Papenburg
- Italy (2):
  - Osp. S. Salvatore, L’Aquila
  - S.Giovanni Bosco, Napoli
- Portugal (3):
  - Hospital Espírito Santo, E.P.E, Evora
  - Hospital Central Faro, Faro
  - Centro Hospitalar Lisboa Norte (CHLN) - Hospital de Santa Maria, Lisbon
- Hospital Universitario Virgen del Rocío, Seville, Spain